CLINICAL TRIAL: NCT00101972
Title: A Phase I, Multi-Dose Study of RAV12 (ANTI-RAAG12 MAB) in Patients With Metastatic or Recurrent Adenocarcinoma
Brief Title: RAV12 in Treating Patients With Metastatic or Recurrent Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000415581; RAVENBIO-RV-2004-002 (Other: Raven biotechnologies (MacroGenics))
Record Dates: First submitted 2005-01-18; First posted 2005-01-19 (Estimated); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Cancer
Keywords: adenocarcinoma of the bladder; adenocarcinoma of the colon; adenocarcinoma of the esophagus; adenocarcinoma of the extrahepatic bile duct; adenocarcinoma of the gallbladder; adenocarcinoma of the lung; adenocarcinoma of the pancreas; adenocarcinoma of the prostate; adenocarcinoma of the rectum; adenocarcinoma of the stomach; adenocarcinoma with squamous metaplasia of the gallbladder; cervical adenocarcinoma; endometrial adenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian undifferentiated adenocarcinoma; salivary gland adenocarcinoma; small intestine adenocarcinoma; vaginal adenocarcinoma; vaginal clear cell adenocarcinoma; ovarian clear cell cystadenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian serous cystadenocarcinoma; stage IV bladder cancer; stage IV breast cancer; stage IV colon cancer; stage IV endometrial carcinoma; stage IV esophageal cancer; stage IV gastric cancer; stage IV non-small cell lung cancer; stage IV ovarian epithelial cancer; stage IV prostate cancer; stage IV rectal cancer; stage IV renal cell cancer; stage IV salivary gland cancer; stage IVA cervical cancer; stage IVA vaginal cancer; stage IVB cervical cancer; stage IVB vaginal cancer; recurrent bladder cancer; recurrent breast cancer; recurrent cervical cancer; recurrent colon cancer; recurrent endometrial carcinoma; recurrent esophageal cancer; recurrent extrahepatic bile duct cancer; recurrent gallbladder cancer; recurrent gastric cancer; recurrent non-small cell lung cancer; recurrent ovarian epithelial cancer; recurrent pancreatic cancer; recurrent prostate cancer; recurrent rectal cancer; recurrent renal cell cancer; recurrent salivary gland cancer; recurrent small intestine cancer; recurrent vaginal cancer; unresectable extrahepatic bile duct cancer; unresectable gallbladder cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms; Adenocarcinoma Of Esophagus; Adenocarcinoma of Lung; Rectal Neoplasms; Urinary Bladder Neoplasms; Breast Neoplasms; Endometrial Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial; Prostatic Neoplasms; Carcinoma, Renal Cell; Salivary Gland Neoplasms; Uterine Cervical Neoplasms; Vaginal Neoplasms; Bile Duct Neoplasms; Gallbladder Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAV12 (Experimental)
  Interventions: Biological: monoclonal antibody RAV12

INTERVENTIONS:
Biological: monoclonal antibody RAV12 — Escalating doses of RAV12 (weekly 0.3, 1.0, 1.5, 3.0, 4.0, 5.0, 6.0 mg/kg or 0.5 mg/kg BIW or TIW; 0.75 mg/kg BIW) for 4 weeks

SUMMARY:
RATIONALE: Monoclonal antibodies, such as RAV12, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

PURPOSE: This phase I trial is studying the side effects and best dose of RAV12 in treating patients with metastatic or recurrent adenocarcinoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of RAV12 in patients with metastatic or recurrent adenocarcinoma.
* Determine the toxicity profile of this drug in these patients.
* Determine the pharmacokinetics and immunogenicity of this drug in these patients.
* Determine, preliminarily, the antitumor activity of this drug in these patients.

OUTLINE: This is an open-label, dose-escalation study.

Patients receive RAV12 IV over 2 hours 2-3 times per week in weeks 1-4 (course 1). Patients are evaluated for response on day 43. Patients achieving a partial or complete response may be eligible to receive additional courses of RAV12 as above. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of RAV12 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Up to 15 additional patients are treated at the MTD in 1 or more patients groups (e.g., colorectal, pancreatic, gastroesophageal, and other adenocarcinoma).

After completion of study treatment, patients are followed within 4 weeks and then every 6-12 months thereafter.

PROJECTED ACCRUAL: A total of 75 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma

  * Metastatic or recurrent disease
  * Not curable by standard therapies
* Must have failed at least 1, but no more than 3, prior therapies for metastatic or recurrent disease

  * Patients with colorectal or breast adenocarcinoma must have failed at least 2 prior therapies
  * Must have had at least stable disease for 3 months while on last treatment prior to most recent disease progression
* Meets 1 of the following criteria:

  * At least 1 measurable site of disease ≥ 2 cm by radiography
  * Evaluable disease that could be reliably and consistently followed, as deemed by the principal investigator
* RAAG12 expression confirmed* by immunohistochemistry NOTE: *Not required for patients with colon, pancreatic, or gastric adenocarcinoma
* No evidence of residual or recurrent CNS metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Not specified

Menopausal status

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* More than 3 months

Hematopoietic

* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL (transfusions allowed)
* Absolute neutrophil count ≥ 1,500/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* γ-glutamyl transferase ≤ 2.5 times ULN
* Adequate hepatic function sufficient to undergo study therapy

Renal

* Creatinine < 1.5 mg/dL
* Adequate renal function sufficient to undergo study therapy

Cardiovascular

* No New York Heart Association class III or IV heart disease
* No thrombosis within the past 3 months, including any of the following:

  * Deep vein thrombosis
  * Myocardial infarction
  * Stroke
* Adequate cardiac function sufficient to undergo study therapy

Pulmonary

* No pulmonary embolism within the past 3 months
* No significant pulmonary compromise, particularly dependence on supplemental oxygen on an as-needed or continuous basis
* Adequate pulmonary function sufficient to undergo study therapy

Immunologic

* No active viral, bacterial or systemic fungal infection requiring parenteral therapy within the past 4 weeks
* No history of chronic or recurrent infection requiring continual antiviral, antifungal, or antibacterial agents
* No known hypersensitivity to murine or recombinant proteins, polysorbate 80, or any excipient contained in study drug

Other

* Amylase and lipase normal
* No other primary malignancy within the past 3 years except for the following:

  * Treated non-melanoma skin cancer
  * Carcinoma in situ of the cervix by biopsy
  * Squamous intraepithelial lesion of the cervix by PAP smear
  * Localized prostate cancer (Gleason score < 6)
  * Resected melanoma in situ
* No other serious medical condition that would preclude study participation
* No dementia or altered mental status that would preclude giving informed consent
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 half-lives since prior monoclonal antibody therapy
* No concurrent vaccinations
* No concurrent prophylactic hematologic growth factors

Chemotherapy

* At least 4 weeks since prior chemotherapy

Endocrine therapy

* No concurrent steroids except for the following:

  * Inhaled, ophthalmic, or nasal steroids
  * Stable dose of oral prednisone (or equivalent) ≤ 10 mg/day

Radiotherapy

* At least 4 weeks since prior radiotherapy

Surgery

* More than 4 weeks since prior major surgery

Other

* More than 4 weeks since prior investigational agents
* Prior oral antiviral, antifungal, or antibacterial therapy allowed provided therapy was completed within the past week
* No other concurrent antineoplastic therapy
* No concurrent immunosuppressive medications
* No other concurrent investigational agents
* No concurrent vitamins except those approved by the medical monitor

  * Concurrent daily multivitamin allowed
* Concurrent bisphosphonates allowed provided patient is on stable dose for ≥ 1 month prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2004-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Toxicity by CTCAE | Days 1-50

SECONDARY OUTCOMES:
Maximum tolerated dose | Days 1-50
Pharmacokinetics of RAV12 by serum levels | Days 1, 2, 4, 5, 8, 15, 22, 29, 36, 43, and 50
Immunogenicity by Human Anti-chimeric antibodies | Days 1, 8, 15, 22, and 50
Time to tumor progression by clinical assessment | 6 months
Progression free survival by clinical assessment | 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Premiere Oncology, Santa Monica, California
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Sarah Cannon Cancer Center at Centennial Medical Center, Nashville, Tennessee

REFERENCES:
- [Result] Burris HA 3rd, Rosen LS, Rocha-Lima CM, Marshall J, Jones S, Cohen RB, Kunkel LA, Loo D, Baughman J, Stewart SJ, Lewis N. Phase 1 experience with an anti-glycotope monoclonal antibody, RAV12, in recurrent adenocarcinoma. Clin Cancer Res. 2010 Mar 1;16(5):1673-81. doi: 10.1158/1078-0432.CCR-09-2263. Epub 2010 Feb 23. PMID 20179219